CLINICAL TRIAL: NCT02619617
Title: A Multicenter, Placebo-Controlled, Single Dose Study in Acute Episodic and Chronic Cluster Headache to Evaluate the Safety and Efficacy of SOM230 Subcutaneous (s.c.)
Brief Title: Safety and Efficacy Study of SOM230 s.c. in Cluster Headache
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Novartis decision based on Cohort 1 results
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: CSOM230Y2201
Record Dates: First submitted 2015-11-30; First posted 2015-12-02 (Estimated); Results first posted 2020-01-13 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2019-12

CONDITIONS: Cluster Headache - Episodic and Chronic
Keywords: Cluster Headache; Patient Diary collection of headache pain
MeSH Terms: conditions — Cluster Headache; Bronchiolitis Obliterans Syndrome | interventions — pasireotide

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- SOM230 0.9mg (Experimental): cohort 2
  Interventions: Drug: SOM230; Drug: Placebo
- SOM230 1.5 mg (Experimental): cohort 1
  Interventions: Drug: SOM230; Drug: Placebo

INTERVENTIONS:
Drug: SOM230 — The study evaluated SOM230 vs Placebo
Drug: Placebo — The study evaluated SOM230 vs Placebo

SUMMARY:
The purpose of this study was to determine if SOM230 is safe and effective for the treament of cluster headache.

DETAILED DESCRIPTION:
The purpose of this non-confirmatory study was to determine if SOM230 has adequate efficacy and safety to warrant further clinical development in cluster headache (CH). This study was a sequential design of SOM230 vs. Placebo.

ELIGIBILITY:
Inclusion Criteria:

* Subject is male or female age 18-65 inclusive.
* Written informed consent must be obtained before any assessment is performed.
* Subjects must have established diagnosis of episodic cluster headaches (CH) or chronic CH, averaging 2-6 headache attacks per day each lasting at least 45 minutes without treatment, not to exceed 6 attacks per day within the last year.
* Able to communicate well with the investigator, to understand and comply with the requirements of the study, as well as accepting NOT to share any study information through social media during their participation in the study.
* Subject is able to self-inject medication subcutaneously or have the assistance of a partner on an out-patient basis.

Exclusion Criteria:

* Subjects that have a history of greater than 6 CH attacks per day within the last year.
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using effective methods of contraception during the duration dosing of the study treatment. Or men who are sexually active with women of child bearing potential, unless the male subjects always use condoms during the study.
* History of multiple and recurring allergies or allergy to the investigational compound/compound class being used in this study.
* Use of other investigational drugs at the time of enrollment, or within 5 half-lives of enrollment, or within 30 days, whichever is longer; or longer if required by local regulations.
* A history of clinically significant heart diseases, ECG abnormalities, continued use of drugs known to prolong QTc during the study conduct, or any of the following ECG abnormalities at screening or baseline:

  * QTcF > 450 msec (males)
  * QTcF > 460 msec (females)
* Uncontrolled diabetes as evidenced by screening HbA1c > 8.0%
* A positive Hepatitis B surface antigen or Hepatitis C test result.
* A positive pregnancy test or lactating mothers.
* History of drug or alcohol abuse within the 12 months prior to dosing other than prescription medications to manage their CH attacks, or evidence of such abuse as indicated by the laboratory assays conducted during screening.
* Significant acute illness which has not resolved within two (2) weeks prior to initial dosing.
* Any surgical or medical condition which might significantly jeopardize the subject's safety in case of participation in the study. The Investigator should make this determination in consideration of the subject's medical history and/or clinical or laboratory evidence of any of the following:
* Liver disease or liver injury as indicated by abnormal liver function tests. ALT (SGPT), AST (SGOT), γ-GT, alkaline phosphatase and serum bilirubin will be tested.
* ALT must be within the normal range
* Serum bilirubin must not exceed 1.2 x ULN
* γ-GT, AST and alkaline phosphatase must not exceed 2 x ULN [If necessary, laboratory testing may be repeated on one occasion (as soon as possible) prior to treatment, to rule out any laboratory error]
* Acute cholecystitis or symptomatic cholelithiasis in subjects without H/O cholecystectomy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2016-10-31 (Actual); Primary Completion 2018-09-25 (Actual); Study Completion 2018-09-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (4):
- United States (2):
  - Novartis Investigative Site, Culver City, California
  - Novartis Investigative Site, Philadelphia, Pennsylvania
- Novartis Investigative Site, Königstein im Taunus, Taunus, Germany
- Novartis Investigative Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- See also: A Plain Language Trial Summary is available on novartisclinicaltrials.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=313

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study was planned to have 2 cohorts using a one-sequence two-period design to compare SOM230 vs. placebo. Two consecutive CH attacks were treated: the first attack was treated with placebo (Period 1) and the subsequent attack was treated with SOM230 (Period 2). However, Cohort 2 was not initiated.
Groups:
- Placebo s.c.: Single dose of placebo
- SOM230 1.5 mg s.c.: Single dose of SOM230 1.5 mg s.c.
Period: Period 1 Placebo - 1st AttacK
Arm/Group | Placebo s.c. | SOM230 1.5 mg s.c.
Started | 28 | 0
Participants Included in PD Analysis | 20 | 0
Participants in Safety Set for Period 1 (participants in Cohort 1 in Period 1 received placebo s.c.) | 28 | 0
Completed | 28 | 0
Not Completed | 0 | 0
Period: Period 2 SOM230 - 2nd Attack
Arm/Group | Placebo s.c. | SOM230 1.5 mg s.c.
Started | 0 | 28
Participants in Safety Set for Period 2 | 0 | 28
Completed | 0 | 24
Not Completed | 0 | 4
Not completed — Protocol Violation | 0 | 1
Not completed — Physician Decision | 0 | 3

BASELINE CHARACTERISTICS:
Population: Safety analysis set excluded 2 subjects due to not being dosed.
Groups:
- Placebo s.c. /1.5 mg SOM230 s.c.: A: single dose of placebo s.c. (Period 1) B: single dose of 1.5 mg s.c. SOM230 (Period 2)
Arm/Group | Placebo s.c. /1.5 mg SOM230 s.c.
Number analyzed (Participants) | 28
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43.9 (10.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 22

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Headache Response (PD Analysis Set)
Description: Defined as very severe, severe, or moderate pain before dosing that becomes mild or nil at 30 minutes post-dosing
Time Frame: 30 minutes post dose
Population: PD analysis set: Subjects with protocol deviations which impacted PD data were excluded from the PD analysis
Measure: Number; unit: participants
Groups:
- Placebo s.c.: A single dose of placebo s.c.
- SOM230 1.5 mg: A single dose of 1.5 mg s.c. SOM230
Arm/Group | Placebo s.c. | SOM230 1.5 mg
Number analyzed (Participants) | 20 | 20
participants | 9 | 10
Statistical Analysis 1: Comparison: Placebo s.c. vs SOM230 1.5 mg; Test type: Other — 1.5mg SOM230 s.c. vs. Placebo s.c; p = 0.698, Regression, Logistic; Odds Ratio (OR) = 1.308, 90% CI 2-sided [0.419 to 4.082]

2. Secondary Outcome: Number of Participants Who Were Pain Free at 30 Minutes Post Dose
Description: Participants who were pain free 30 minutes after dosing and reporting improvement of associated autonomic symptoms (for example, lacrimation, blushing, pupil constriction, etc.) over time was tabulated by dose.
Time Frame: 30 mins post dose
Population: PD analysis set)
Measure: Number; unit: participants
Groups:
- SOM230 1.5 mg: single dose of 1.5 mg s.c. SOM230
Arm/Group | Placebo s.c. | SOM230 1.5 mg
Number analyzed (Participants) | 20 | 20
participants | 5 | 7
Statistical Analysis 1: Comparison: Placebo s.c. vs SOM230 1.5 mg; Test type: Other — 1.5mg SOM230 s.c. vs. Placebo s.c; p = 0.385, Regression, Logistic; Odds Ratio (OR) = 2.033, 90% CI 2-sided [0.530 to 7.790]

3. Secondary Outcome: Change in Hemoglobin Values From Screening to End of Study
Description: Change in hemoglobin values from screening and end of study
Time Frame: screening and end of study, up to 9 days after treatment
Population: Safety analysis set
Measure: Mean (Standard Deviation); unit: g/L
Groups:
- Placebo s.c. /1.5 mg SOM230 s.c.: A: single dose of placebo s.c. B: single dose of 1.5 mg s.c. SOM230
Arm/Group | Placebo s.c. /1.5 mg SOM230 s.c.
Number analyzed (Participants) | 28
g/L
  Screening | 153.4 (12.93)
  End of Study | 149.5 (15.13)

4. Secondary Outcome: Pulse Rate
Description: Vital signs by treatment and time point
Time Frame: screening and end of study, up to 9 days after treatment
Population: Safety analysis set
Measure: Mean (Standard Deviation); unit: Beats/min
Arm/Group | Placebo s.c. /1.5 mg SOM230 s.c.
Number analyzed (Participants) | 28
Beats/min
  Screening | 77.2 (15.02)
  Baseline | 78.1 (11.99)
  Period 1 - Placebo: number analyzed (Participants) | 17
  Period 1 - Placebo | 76.9 (12.77)
  Period 2 - SOM230 1.5 mg: number analyzed (Participants) | 24
  Period 2 - SOM230 1.5 mg | 74.0 (10.86)
  End of Study: number analyzed (Participants) | 27
  End of Study | 81.1 (13.50)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from first dose of study treatment until end of study treatment plus 30 days post treatment, up to maximum duration of 26 months.
Groups:
- 1.5 mg SOM230 s.c.: single dose of 1.5 mg s.c. SOM230
Arm/Group | 1.5 mg SOM230 s.c. | Placebo s.c.
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/28
Other Adverse Events (participants affected / at risk) | 23/26 | 5/28
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 1.5 mg SOM230 s.c. (N=26) | Placebo s.c. (N=28)
Palpitations (Cardiac disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 0
Diarrhoea (Gastrointestinal disorders) | 7 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 12 | 0
Vomiting (Gastrointestinal disorders) | 7 | 1
Fatigue (General disorders) | 6 | 1
Injection site bruising (General disorders) | 0 | 1
Injection site erythema (General disorders) | 4 | 1
Injection site pain (General disorders) | 5 | 1
Injection site reaction (General disorders) | 1 | 1
Injection site warmth (General disorders) | 1 | 0
Malaise (General disorders) | 1 | 0
Vessel puncture site bruise (General disorders) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0
Haematocrit decreased (Investigations) | 1 | 0
Red blood cell count decreased (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 0
Dizziness (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 2 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Flushing (Vascular disorders) | 1 | 1

LIMITATIONS AND CAVEATS:
Terminated (Non-efficacy in first Phase 2a cohort.)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2018-03-14): https://cdn.clinicaltrials.gov/large-docs/17/NCT02619617/Prot_000.pdf
  • Statistical Analysis Plan (2018-11-09): https://cdn.clinicaltrials.gov/large-docs/17/NCT02619617/SAP_001.pdf